CLINICAL TRIAL: NCT02384239
Title: Palbociclib in Combination With Fulvestrant or Tamoxifen as Treatment for Hormone Receptor Positive Metastatic Breast Cancer Previously Exposed to Inhibitors of the PI3K Pathway: A Phase II Study With Pharmacodynamics Markers
Brief Title: A Study of Palbociclib in Combination With Fulvestrant or Tamoxifen as Treatment for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Hope Rugo, MD, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147522; NCI-2015-01791 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2015-02-10; First posted 2015-03-10 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Breast Cancer; Hormone Receptor Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Tamoxifen; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Palbociclib 100mg and, fulvestrant or tamoxifen (Experimental): Palbociclib dose 100mg, and either fulvestrant (500 mg IM on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
  Interventions: Drug: Palbociclib; Drug: Tamoxifen; Drug: Fulvestrant
- Palbociclib 125mg and, fulvestrant or tamoxifen (Experimental): Palbociclib dose 125mg and either fulvestrant (500 mg IM on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
  Interventions: Drug: Palbociclib; Drug: Tamoxifen; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Given orally (PO)
  Other Names: Ibrance
Drug: Tamoxifen — Given orally (PO)
  Other Names: Tamoxifen 20mg
Drug: Fulvestrant — Given by intramuscular (IM) injection.
  Other Names: Faslodex

SUMMARY:
This phase II trial studies the side effects of palbociclib when given together with fulvestrant or tamoxifen citrate in treating patients with hormone receptor positive breast cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or has spread to other places in the body (metastatic). Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hormone therapy using fulvestrant or tamoxifen citrate may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving palbociclib together with fulvestrant or tamoxifen citrate may work better in treating hormone receptor positive breast cancer.

DETAILED DESCRIPTION:
Patients will be randomly allocated in a 1:1 ratio to take either 100 mg or 125 mg of palbociclib. Randomized treatment assignments will be made by permuted blocks, generated by our collaborating statistician at Dana-Farber Cancer Institute.

PRIMARY OBJECTIVES:

I. To evaluate the incidence of grade 3/4 neutropenia in patients with hormone receptor positive (HR+) advanced breast cancer previously exposed to chemotherapy, treated with fulvestrant or tamoxifen (tamoxifen citrate) in combination with palbociclib at a dose of 100mg or 125mg.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival with 100 mg and 125 mg dosing of palbociclib.

II. To evaluate inhibition of retinoblastoma (RB) phosphorylation in tumor and in skin at 100 mg and 125 mg dosing of palbociclib.

III. To evaluate the correlation between inhibition of RB phosphorylation in skin and tumor.

IV. To evaluate the correlation between inhibition of RB phosphorylation and progression-free survival (PFS).

V. To evaluate the objective response and clinical benefit rate of palbociclib given at 100 mg or 125 mg.

VI. To evaluate the toxicity associated with palbociclib given at 100 mg and 125 mg in combination with fulvestrant or tamoxifen.

VII. To evaluate markers of resistance to palbociclib and fulvestrant or tamoxifen in circulating plasma tumor deoxyribonucleic acid (DNA) (ptDNA).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive low-dose palbociclib orally (PO) on days 1-21. Patients also receive tamoxifen citrate PO on days 1-28 or fulvestrant intramuscularly (IM) on days 1 and 15 of cycle 1 and then on day 1 only in subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive high-dose palbociclib PO on days 1-21. Patients also receive tamoxifen citrate PO on days 1-28 or fulvestrant IM on days 1 and 15 of cycle 1 and then on day 1 only in subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer with evidence of metastatic or locally advanced disease, not amenable to resection or radiation therapy with curative intent.
* Patients 18 years of age or older, Female patients should be either:
* Postmenopausal, as defined by at least one of the following criteria:
* Age >=60 years;
* Age <60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause;
* Documented bilateral oophorectomy;
* Medically confirmed ovarian failure.

OR

* Pre/peri-menopausal, ie, not meeting the criteria for being postmenopausal who are also receiving ongoing treatment with Luteinizing hormone-releasing hormone (LHRH) agonists (goserelin or leuprolide). The first injection should occur at least two weeks before study start.
* Documentation of ER-positive and/or PR-positive tumor (≥1% positive stained cells) based on most recent tumor biopsy (unless bone-only disease,discuss with study PI if results are discordant) utilizing an assay consistent with local standards.
* Documented human epidermal growth factor receptor 2 negative (HER2-) tumor based on local testing on most recent tumor biopsy: HER2-negative tumor is determined as immunohistochemistry score 0/1+ or negative by in situ hybridization (FISH/CISH/SISH) defined as a HER2/CEP17 ratio <2 or for single probe assessment a HER2 copy number <4.
* Must have received prior treatment with an Mechanistic target of rapamycin (mTOR) or phosphatidylinositol 3-kinase (PI3K) inhibitor
* Up to 2 prior lines of chemotherapy are allowed in the metastatic setting.
* Any number of lines of prior hormone therapy are allowed
* Patients with clear progression on either tamoxifen or fulvestrant should receive the alternate agent. Patients with clear progression on both drugs are not eligible.
* Ability to have a skin and tumor biopsy. Patients without accessible tumor for biopsy will be considered on a case by case basis.
* Patients who cannot be biopsied will not be replaced (although up to 5 ineligible/inevaluable patients can be replaced)
* A patient without biopsy amenable tumor must be cleared by the PI of the study; up to 10 patients without biopsy amenable tumor will be allowed in each arm of the study.
* Patients without accessible tumor for biopsy must provide archived tumor from the most recent biopsy available
* Bone marrow, hepatic, and renal function as follows:

Adequate bone marrow function:

* leukocytes > 2500/mL
* absolute neutrophil count > 1,000/mL
* platelets > 100,000/mL"

Adequate hepatic function:

* total bilirubin within normal institutional limits (unless Gilbert's disease with elevated indirect bilirubin only)
* aspartate aminotransferase (AST) / (serum glutamic-oxaloacetic transaminase (SGOT) < 2.5 X institutional upper limit of normal
* alanine aminotransferase (ALT) / (serum glutamic-pyruvic transaminase (SGPT) < 2.5 X institutional upper limit of normal
* Adequate renal function:
* creatinine within normal institutional limits
* Measurable or evaluable disease as defined by RECIST version 1.1. Tumor lesions previously irradiated or subjected to other loco-regional therapy will only be deemed measurable if progression at the treated site after completion of therapy is clearly documented.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Resolution of acute toxic effects of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE Grade <=1 (except alopecia)
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Prior treatment with any cyclin-dependent kinase (CDK) inhibitor, and/or both fulvestrant and tamoxifen in the metastatic setting with clear progression.
* Patients with advanced/metastatic, symptomatic, visceral spread, at risk of life-threatening complications in the short term by investigator assessment.
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated (eg, radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization .
* Current use of food or drugs known to be potent CYP3A4 inhibitors, drugs known to be potent CYP3A4 inducers (for examples, see the prohibited medications section), and drugs that are known to prolong the QT interval. See prohibited meds in appendix 5.
* Major surgery, chemotherapy, radiotherapy, or other anti-cancer therapy within 2 weeks before randomization.
* Any other malignancy within 3 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* QTc interval >480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.

QTc (Bazett) = QT/√RR

* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, symptomatic congestive heart failure, or cerebrovascular accident excluding transient ischemic attack.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of palbociclib, such as history of GI surgery with may result in intestinal blind loops and patients with clinically significant gastroparesis, short bowel syndrome, unresolved nausea, vomiting, active inflammatory bowel disease or diarrhea of CTCAE v4.0 Grade >1.
* Prior hematopoietic stem cell or bone marrow transplantation.
* Abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants (that cannot be safely held for biopsy) that would preclude tumor and skin biopsies.
* For fulvestrant: Ongoing anticoagulation that would preclude an IM injection
* For tamoxifen: Documented hypercoagulable state not receiving anticoagulation
* Known or possible hypersensitivity to palbociclib (CTCAE v4.0).
* Known human immunodeficiency virus infection.
* Other severe acute or chronic medical or psychiatric condition, including recent or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Participation in other studies involving investigational drug(s) (Phases 1-4) within 2 weeks before randomization the current study.
* Women should not become pregnant or breastfeed whilst on this study. Birth control methods are acceptable and will be discussed with study participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Palbociclib 100mg: Palbociclib dose 100mg, and either fulvestrant (500 mg intramuscular injection (IM) on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
- Palbociclib 125mg: Palbociclib dose 125mg and either fulvestrant (500 mg IM on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
Period: Overall Study
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Palbociclib 100mg: Palbociclib dose 100mg, and either fulvestrant (500 mg IM on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
- Total: Total of all reporting groups
Arm/Group | Palbociclib 100mg | Palbociclib 125mg | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 0 | 1
  40-49 years old | 5 | 7 | 12
  50-59 years old | 11 | 15 | 26
  60-69 years old | 12 | 5 | 17
  70-79 years old | 5 | 6 | 11
  80-89 years old | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 1 | 3
  White | 28 | 26 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or 4 Neutropenia
Description: Grade 3/4 neutropenia as defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.03 in patients with prior exposure to 1-3 lines of chemotherapy for metastatic breast cancer
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 34
percentage of participants | 19.4 | 20.5

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as the interval from study entry to the first documented evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as at least a 20% increase in the sum of the longest diameter (SLD) of target lesions, taking as reference the smallest sum SLD recorded since the treatment started and minimum 5 mm increase over the nadir, or the appearance of one or more new lesions. Patients who remain progression-free at the time of analysis will be censored at their last date of follow-up.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 34
months | 6.53 [2.33 to 12.2] | 9.4 [3.56 to 19.7]

3. Secondary Outcome: Proportion of Participants With Demonstrated Clinical Benefit
Description: Defined as the proportion of patients whose best overall response, according to RECIST, is either complete response (CR), a partial response (PR) or stable disease (SD) at 24 weeks. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Time Frame: 24 weeks
Population: Two participants in the 125mg group did not have an evaluable disease assessment 24 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 32
proportion of participants | 0.67 | 0.75

4. Secondary Outcome: Proportion of Participants With an Objective Response
Description: Defined as the proportion of patients whose best overall response, according to RECIST, is either complete response (CR), a partial response (PR) at 24 weeks. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Time Frame: 24 weeks
Population: Two participants in the 125mg group did not have an evaluable disease assessment 24 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 32
proportion of participants | 0.1111 | 0.0625

5. Secondary Outcome: Median Change in Percent Positive Cells From Baseline of Ki-67
Description: Median change in percent positive cells of Ki-67 from baseline will be reported with IQR
Time Frame: Up to 24 months
Measure: Median (Inter-Quartile Range); unit: change in percent positive cells
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 34
change in percent positive cells | -8 [-22 to 0] | -6 [-19 to -1]

6. Secondary Outcome: Median Change in Percent Positive Cells From Baseline of Total-Rb
Description: Median change in percent positive cells of Total-Rb from baseline will be reported with interquartile range (IQR)
Time Frame: Up to 24 months
Measure: Median (Inter-Quartile Range); unit: change in percent positive cells
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 34
change in percent positive cells | 4 [-25 to 30] | 5 [-15 to 29]

7. Secondary Outcome: Median Change in Percent Positive Cells From Baseline of pS780-Rb
Description: Median change in percent positive cells of pS780-Rb from baseline will be reported with IQR
Time Frame: Up to 24 months
Measure: Median (Inter-Quartile Range); unit: change in percent positive cells
Groups:
- Palbociclib 100mg: Treatment arm palbociclib dose 100mg + fulvestrant or tamoxifen
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
Number analyzed (Participants) | 36 | 34
change in percent positive cells | -3 [-32 to 4] | -6 [-14 to 12]

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- Palbociclib 100mg: Palbociclib dose 100mg and either fulvestrant (500 mg IM on days 1 and 15 in the first 28 days, then every 28 days thereafter) or tamoxifen (20 mg PO daily by physician choice)
Arm/Group | Palbociclib 100mg | Palbociclib 125mg
All-Cause Mortality (participants affected / at risk) | 3/36 | 1/34
Serious Adverse Events (participants affected / at risk) | 5/36 | 2/34
Other Adverse Events (participants affected / at risk) | 7/36 | 9/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib 100mg (N=36) | Palbociclib 125mg (N=34)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib 100mg (N=36) | Palbociclib 125mg (N=34)
Neutrophil count decreased (Investigations) | 5 (12) | 9 (19)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT02384239/Prot_SAP_000.pdf